CLINICAL TRIAL: NCT02634775
Title: Part 3 of: 'Conceptualisation and Validation of a Paradigm Based on Uraemic Toxins for Management of Chronic Kidney Disease in Paediatric Patients (UToPaed)'
Brief Title: Uraemic Toxins in Chronic Kidney Disease Paediatric Patients: Interventional Study
Acronym: UToPaed_3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UGent_UToPaed_3
Record Dates: First submitted 2015-12-01; First posted 2015-12-18 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Disease
Keywords: Pediatrics; Nephrology; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CKD - no dialysis (Experimental): Change in treatment strategy: Start on dialysis, transplantation
  Interventions: Other: Change in treatment strategy
- Patients on PD (Experimental): Change in treatment strategy: Change of PD prescription, start on HD, transplantation
  Interventions: Other: Change in treatment strategy
- Patients on HD (Experimental): Change in treatment strategy: Change of HD prescription, transplantation
  Interventions: Other: Change in treatment strategy

INTERVENTIONS:
Other: Change in treatment strategy — Start on dialysis, transplantation, change of PD prescription, change of HD prescription

SUMMARY:
Children with chronic kidney disease (CKD) suffer from one of the most devastating diseases in childhood resulting in a lifelong need for health care, and a 3 times decreased life expectancy. In addition, they have important comorbidities that negatively impact on their quality of life and integration in society, jeopardizing their future even after a potential transplantation. Retention of uraemic toxins is accepted to play a major role in the pathogenesis of the comorbid conditions, but studies in children are lacking. Furthermore, there are currently no good tools to evaluate severity and monitor adequacy of treatment, resulting in suboptimal management.

The overall scientific objective of this four years UToPaed IWT-TBM project is to provide the clinician with new diagnostic and therapeutic tools for the management of children with CKD, based on the improved understanding of uraemic toxicity.

In UToPaed (part 1), the investigators will associate concentrations of a wide variety of uraemic toxins with different comorbidities in CKD children, i.e. growth, protein-energy wasting, quality of life, cardiovascular risk factors, circadian rhythm, sleep quality, and psychosocial and neurocognitive functioning (i.e. cross-sectional and longitudinal). Those toxins of which concentrations are best correlated with comorbidities during the progress of CKD and those having representative kinetics (UToPaed - part 2: Kinetic analysis) will be selected as markers. During this third part of UToPaed, these markers will be, together with the comorbidities, further tracked after interventions, i.e. starting on dialysis, transplantation, changes in dialysis strategy.

From the validated kinetic models (UToPaed - part 2 and 3), an open access user-friendly prediction simulator (PAEDSIM) based on patient characteristics and marker concentrations will be developed to optimise and individualise the dialysis therapy.

By providing clinicians with more advanced and appropriate tools to improve management of all children with CKD, i.e. better assessment of the degree of renal dysfunction, better determination of the ideal time to start renal replacement therapy, and more accurate monitoring of dialysis adequacy, the investigators aim to improve neurocognitive and psychosocial functioning (short term), growth, maturation into puberty, and social integration (median term) and survival (long term).

DETAILED DESCRIPTION:
This is an interventional multicenter study in children (≤ 18 years) with chronic kidney disease (CKD) stage 2 to 5D with or without renal replacement therapy. They will be followed for a total duration of 24 months.

Concentrations of the uraemic toxin markers and the different comorbidities will be followed after an intervention. Some interventions will just happen in the treatment of the CKD child: e.g. transplantation, start on dialysis, needed switch from PD to HD.

In the patients on PD, different approaches will be followed: more frequent exchanges overnight, PET-directed dialysis regimes, adapted PD, using a mix of short, small volume dwells, with longer, high volume dwells. These different strategies have so far only been tested using the classic adequacy parameters urea and creatinine. The intervention is that the children, as included in the longitudinal study, will be studied while on at least two different PD strategies, serving as their own control, whereby the strategy will be linked with the concentration of the uraemic toxin markers and comorbidities.

In the patients on HD, different dialysis strategies will be studied: conventional haemodialysis 3x/week, daily haemodialysis, haemodiafiltration 3x/week, nocturnal 8h dialysis 3x/week, and the optimal dialysis regime as derived from the kinetic analysis (UToPaed_2). The intervention is that the children, as included in the longitudinal study, will be studied with at least 2 of the strategies, and that differences in plasma concentrations and removal rate of the uraemic toxin markers will be measured. The measured predialysis concentrations, time averaged concentrations (TACs), and total solute removal with the different strategies will be compared to the results of the kinetic simulations in order to validate the calibrated kinetic models of the uraemic toxin markers.

Based on the results, guidance on the most optimal dialysis strategy for each child will be developed, and the child will consequently be treated on that modality during 1 year, to allow evaluation of the longer term impact on quality of life, catch up growth, study results and emergence of new comorbidities.

The therapeutic tool comprises an open access user-friendly prediction simulator, based on the kinetics of the new markers (PAEDSIM) to simulate different dialysis strategies. With different patient characteristics and uraemic toxin concentrations as input for the simulation model, the program will derive the optimal dialysis strategy for the individual patient striving for low predialysis concentrations and TACs.

The clinical use of these findings will be promoted by the organisation of a 'CKD Academy' with workshops about the prediction simulator (PAEDSIM) and the related laboratory techniques (see utilisation strategies).

ELIGIBILITY:
Subject Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged ≤ 18 years
* Diagnosed with chronic kidney disease stage 2 to 5D, according to the K/DOQI guidelines.

Subject Exclusion Criteria:

* N.A.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of concentrations of uraemic toxins as measured in HD patients after interventions with those as will be predicted by the kinetic model (model validation) | up to 4 years

SECONDARY OUTCOMES:
Decrease of blood concentrations of uraemic toxins in PD and HD patients by changing dialysis prescription to the optimal dialysis strategy | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Eloot, Prof Dr, Principal Investigator — Ghent University Hospital - Nephrology; Johan Vande Walle, Prof Dr, Study Chair — Ghent University Hospital - Paediatric Nephrology; Ann Raes, Prof Dr, Study Chair — Ghent University Hospital - Paediatric Nephrology; Wim Van Biesen, Prof Dr, Study Chair — Ghent University Hospital - Nephrology; Evelien Snauwaert, Study Chair — Ghent University Hospital - Paediatric Nephrology
Locations (1):
- Ghent University Hospital - Nephrology, Ghent, Belgium